CLINICAL TRIAL: NCT03387683
Title: A Double-blind, Randomized, Parallel Group, Phase IV Study to Investigate the Effects of DAPAgliflozin on CARDiac Substrate Uptake, Myocardial Efficiency and Myocardial Contractile Work in Type 2 Diabetes Patients
Brief Title: A Clinical Study to Investigate the Effects of Dapagliflozin on Heart Work, Heart Nutrient Uptake, and Heart Muscle Efficiency in Type 2 Diabetes Patients
Acronym: DAPACARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1690C00063; 2017-003820-58 (EudraCT Number)
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo tablets once daily
  Interventions: Drug: placebo
- dapagliflozin 10mg (Experimental): dapagliflozin 10mg tablets once daily
  Interventions: Drug: dapagliflozin

INTERVENTIONS:
Drug: dapagliflozin — dapagliflozin 10mg
  Other Names: Forxiga 10mg
  Arms: dapagliflozin 10mg
Drug: placebo — placebo to match dapagliflozin
  Arms: placebo

SUMMARY:
This is a randomised, placebo-controlled, double-blind, parallel-group, international, multicentre, Phase IV study to investigate the effects of dapagliflozin on cardiac substrate uptake, myocardial efficiency and myocardial contractile work in T2D patients. Eligible subjects with T2D before randomisation and fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomised in a 1:1 ratio to dapagliflozin 10 mg or placebo once daily and treated for six weeks. The study includes five visits.

DETAILED DESCRIPTION:
The following will be assessed at Baseline and at the end of the treatment period;

1. MRI scanning in order to assess cardiac function and morphology. The MRI scanning will be made after fasting for at least 6 hours in the same time of day at all visits. The cardiac MRI examination will be performed in accordance with a pre-defined MRI protocol, with the total scan time at each visit estimated to 45 minutes. Images from all sites will be analyzed centrally at the core-lab using a dedicated software package and certified analysts.
2. CT-PET scanning will be made to assess myocardial function and metabolism, as well as fatty acid metabolism in brain, liver and kidney cortex. The CT-PET scanning will be made after a fast as well as abstinence from nicotine, alcohol and caffeine for at least 6 hours at the same time of day at all visits.

   * A cardiac 11C-Acetate PET/CT examination is performed (IV 400 MBq 11C-Acetate).
   * A cardiac 18F-FTHA PET/CT examination is performed (IV 150 MBq 18F-FTHA). The subject is further examined by PET/CT over the liver, kidney cortex and brain (in this order) for uptake of 18F-FTHA. Arterialized venous samples are acquired throughout to assess P-NEFA and 18F-FTHA metabolism by metabolite analysis

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
* Females or males ≥40 years up to 75 years of age.
* Individuals with type 2 diabetes diagnosed for at least 6 months based on the American Diabetes Association standards (ADA, 2017) and on stable dose of metformin for at least 6 weeks prior to screening and HbA1c at screening visit of ≥42 mmol/mol (6.0%) and ≤75 mmol/mol (9.0%) measured at local hospital laboratory.
* No significant signs or symptoms of coronary artery disease or, if known coronary artery disease, currently free of symptoms and a) all major epicardial vessels with <50% stenosis within 12 months prior to screening, or b) if revascularized with all major epicardial vessels with <50% remaining stenosis after stenting or bypass surgery procedure determined between 3 and 12 months prior to screening.
* Normal left ventricular ejection fraction (≥50%) assessed within 1 year prior to informed consent, and if applicable, after most recent acute episode of coronary artery syndrome, or at screening visit.
* Body mass index (BMI) ≥ 25 kg/m2.

Exclusion Criteria:

* Blood pressure at screening that would require a change in blood pressure treatment over the study period or any of the following: systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg.
* History of stroke or other clinically significant cerebrovascular disease.
* Any of the following cardiovascular diseases known within 3 months prior to signing the consent at enrolment:

  1. Atrial fibrillation, or other unstable or severe arrhythmia affecting heart function
  2. Unstable heart failure or any heart failure with NYHA class III and IV
  3. Significant valvular disease
  4. Significant peripheral artery disease
* Planned cardiac surgery or angioplasty within 3 months from enrolment.
* Clinical diagnosis of type 1 diabetes, maturity onset diabetes of the young (MODY), secondary diabetes or diabetes insipidus.
* Verified body weight variability of >3 kg during the 3 proceeding months before screening.
* Active malignancy requiring treatment at the time of visit 1 (with the exception of successfully treated basal cell or treated squamous cell carcinoma).
* Patients with severe hepatic impairment (Child-Pugh class C).
* Unstable or rapidly progressing renal disease.
* Clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Ongoing treatment with other antidiabetic drugs than metformin.
* Ongoing treatment with loop diuretics.
* Ongoing weight-loss diet (hypocaloric diet) or use of weight loss agents.
* Contraindications to dapagliflozin therapy.
* Ongoing treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except for T2D.
* Previous enrolment in the present study or participation in another clinical study with an investigational product during the last 1 month prior to screening.
* Estimated Glomerular Filtration Rate (eGFR) <45 mL/min/1.73 m2.
* Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study treatment intake.
* Any condition when MRI and CT-PET is contraindicated such as, but not limited to, having a metallic implant (such as pacemaker or cochlear implant), permanent make up, claustrophobia or BMI ≥40 kg/m2).
* Involvement in the planning and/or conduct of the study.
* Plasma donation within one month of screening or any blood donation/blood loss >450 mL during the 3 months prior to screening.
* Women who has a positive pregnancy test at enrolment or randomization, or are breastfeeding.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Oldgren, MD, PhD, Principal Investigator — Uppsala Clinical Research Center, Upppsala Sweden; Pirjo Nuutila, MD, PhD, Principal Investigator — University of Turku, Turku, Finland
Locations (2):
- Research Site, Turku, Finland
- Research Site, Uppsala, Sweden

REFERENCES:
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00063&attachmentIdentifier=fab41a7e-3728-4449-af49-b295cc99007e&fileName=D1690c00063-redacted_SAP_-Final_from_PRS.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00063&attachmentIdentifier=bb010979-d9fe-4e2f-bf31-506b76fa8ffa&fileName=D1690C00063-redacted_CSP_from_PRS.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty three patients with type 2 diabetes and on a stable dose of metformin for at least 6 weeks were enrolled in 1 study center in Sweden and 1 center in Finland. The first patient was enrolled on 28 February 2018 and the last patient's last visit was on 19 March 2019.
Pre-assignment Details: Eligible patients were aged between 40 and 75 years, had type 2 diabetes for at least 6 months and had no significant coronary artery disease symptoms. Patients were randomized in a 1:1 ratio, to receive 10 milligram (mg) dapagliflozin or placebo.
Groups:
- Dapagliflozin 10 mg: Patients were randomized to receive an oral dose of 10 mg dapagliflozin, once daily, for 6 weeks.
- Placebo: Patients were randomized to receive an oral dose of placebo (to match 10 mg dapagliflozin), once daily, for 6 weeks.
Period: Overall Study
Arm/Group | Dapagliflozin 10 mg | Placebo
Started | 27 | 26
Completed | 25 | 26
Not Completed | 2 | 0
Not completed — In receipt of disallowed medication | 1 | 0
Not completed — Did not receive treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10 mg | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 12 | 11 | 23
  ≥65 years | 15 | 15 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 19 | 11 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Global Longitudinal Strain of the Left Ventricle (GLSLV) at End of Treatment.
Description: Patients underwent magnetic resonance imaging (MRI) examination to determine the GLSLV, which is expressed as a percentage. The least square mean (LSM) change from baseline estimates were generated from an analysis of covariance (ANCOVA) model with treatment and baseline value of the endpoint as covariates.
Time Frame: Baseline (Day 1) and end of treatment (Day 42)
Population: Patients in the MRI evaluable analysis set who, as per clinical judgment, had fasted and abstained from products containing nicotine, caffeine and alcohol for at least 6 hours prior to both of the times when MRI measurements were taken.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of GLSLV
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of GLSLV | 0.30769 [-0.35001 to 0.96538] | -0.00352 [-0.66121 to 0.65417]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Difference in LSM (Placebo-Dapagliflozin 10 mg); Test type: Other; p = 0.504, ANCOVA — Statistical significance was inferred at a (2-sided) 0.05 level; The LSM estimate and corresponding p-value were obtained from a linear model with treatment and baseline value of the endpoint as covariates; Difference in LSM = 0.31121, 95% CI 2-sided [-0.61900 to 1.24141], Standard Error of Mean 0.46184

2. Secondary Outcome: Adjusted Mean Change From Baseline in Myocardial Efficiency at End of Treatment.
Description: A clinical radiologic assessment of acquired computed tomography and positron emission tomography (CTPET)-[11C]-acetate images was performed to determine myocardial efficiency. The myocardial efficiency calculation was based on an estimate of energy used for producing LV contractile work (mean arterial pressure (MAP) x stroke volume (SV) x heart rate (HR) / myocardial mass) compared to the total cardiac work (calculated based on the total myocardial oxygen consumption per myocardial mass) and is expressed as a percentage. The LSM change from baseline estimates, were generated from an ANCOVA model with treatment and baseline value of the endpoint as covariates.
Time Frame: Baseline (Day 1) and end of treatment (Day 42)
Population: Patients in the CTPET-[11C]-acetate evaluable analysis set who, as per clinical judgment, had fasted and abstained from products containing nicotine, caffeine and alcohol for at least 6 hours prior to both of the times when CTPET-[11C]-acetate measurements were taken.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Myocardial Efficiency
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
Percentage of Myocardial Efficiency | -0.71474 [-3.74654 to 2.31706] | -2.46443 [-5.49623 to 0.56737]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Difference in LSM (Placebo - Dapagliflozin 10 mg); Test type: Other; p = 0.427, ANCOVA — Statistical significance was inferred at a (2-sided) 0.05 level; [statistical method as in outcome 1, analysis 1]; Difference in LSM = 1.74969, 95% CI 2-sided [-2.64837 to 6.14775], Standard Error of Mean 2.18363

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from start of treatment until 1 week after end of treatment (Day 1 to Day 49).
Description: Collection of AE data was limited to the collection of Serious AEs and AEs leading to the discontinuation of study medication only. Data is presented for the Safety Analysis Set which consisted of all subjects who received at least one dose of study medication during the treatment period.
Arm/Group | Dapagliflozin 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03387683/SAP_000.pdf
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03387683/Prot_001.pdf